CLINICAL TRIAL: NCT00860665
Title: Case Volume and Adenoma Detection Rates During Screening Colonoscopy
Brief Title: Case Volume and Adenoma Rate During Screening Colonoscopy
Status: Completed | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Interest group of Berlin private practice gastroenterologists (Unknown)
Responsible Party: Prof. Dr. Thomas Rösch, Department of Interdisciplinary Endoscopy, University Hospital Hamburg Eppendorf, Germany
Other Study IDs: BECOP-3
Record Dates: First submitted 2009-03-11; First posted 2009-03-12 (Estimated); Last update posted 2009-03-12 (Estimated); Status verified 2009-03

CONDITIONS: Colorectal Cancer
Keywords: colorectal cancer; prevention; colonoscopy; screening; quality assessment; colorectal cancer prevention
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Observational study on consecutive persons over the age of 55 years presenting for screening colonoscopy

SUMMARY:
Screening colonoscopy has been established as the most effective means of colorectal cancer prevention. This is based on the fact that colonoscopy detects and removes colonic polyps (adenomas) which are known to progress to cancer if left untreated. The present study examines the question whether case volume (i.e., the number of colonoscopies performed per year) correlates with colonoscopy quality, i.e., adenoma detection rate.

DETAILED DESCRIPTION:
21 private practice gastroenterologist endoscopists from Berlin performed a prospective quality assessment study including at least 10.000 screening colonoscopies. After informed consent, patients data are included (age, sex, family history, colonoscopy performance parameters and findings, therapy performed, histology of biopsies and/or polypectomies, complications (immediate and late) and patient acceptance. The latter was retrieved by patient questionnaires returned after a minimum of 2 weeks. Data were centrally collected in an anonymized way

Primary outcome parameter:

* Correlation of adenoma detection rate with case volume and other confounding factors (e.g., withdrawal time)

Secondary outcome parameters:

* Complications and method of assessment (immediate recording versus later questionnaire enquiry)
* Quality of bowel preparation in relation to outcome Patient acceptance in relation to procedural factors (e.g., sedation)
* Quality of pathology reports and histologic outcome of polypectomy

Later follow-up (after 5-10 years) of the preventive effect of colonoscopy is planned and has been part of the protocol and patient consent form.

ELIGIBILITY:
Inclusion Criteria:

* all persons willing and able to undergo screening colonoscopy over the age of 55 years

Exclusion Criteria:

* any condition not compatible with the definition of screening colonoscopy

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In Germany screening colonoscopy is reimbursed over the age of 55 years. All persons willing to undergo screening colonsocopy without contraindications are asked for consent to be included
Sampling Method: Non-Probability Sample
Enrollment: 12134 (Actual)
Dates: Start 2006-10; Primary Completion 2008-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Correlation of adenoma detection rate with case volume of endoscopists | 18 months

SECONDARY OUTCOMES:
Patient acceptance in relation to procedural factors (e.g. sedation) | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Rösch, MD, Principal Investigator — Department of Interdisciplinary Endoscopy, Hamburg University Eppendorf, Germany
Locations (1):
- Charité Medical University Berlin Campus Virchow, Berlin, State of Berlin, Germany

REFERENCES:
- [Derived] Adler A, Lieberman D, Aminalai A, Aschenbeck J, Drossel R, Mayr M, Mross M, Scheel M, Schroder A, Keining C, Stange G, Wiedenmann B, Gauger U, Altenhofen L, Rosch T. Data quality of the German screening colonoscopy registry. Endoscopy. 2013 Oct;45(10):813-8. doi: 10.1055/s-0033-1344583. Epub 2013 Sep 9. PMID 24019130
- [Derived] Adler A, Wegscheider K, Lieberman D, Aminalai A, Aschenbeck J, Drossel R, Mayr M, Mross M, Scheel M, Schroder A, Gerber K, Stange G, Roll S, Gauger U, Wiedenmann B, Altenhofen L, Rosch T. Factors determining the quality of screening colonoscopy: a prospective study on adenoma detection rates, from 12,134 examinations (Berlin colonoscopy project 3, BECOP-3). Gut. 2013 Feb;62(2):236-41. doi: 10.1136/gutjnl-2011-300167. Epub 2012 Mar 22. PMID 22442161
- [Derived] Adler A, Aminalai A, Aschenbeck J, Drossel R, Mayr M, Scheel M, Schroder A, Yenerim T, Wiedenmann B, Gauger U, Roll S, Rosch T. Latest generation, wide-angle, high-definition colonoscopes increase adenoma detection rate. Clin Gastroenterol Hepatol. 2012 Feb;10(2):155-9. doi: 10.1016/j.cgh.2011.10.026. Epub 2011 Nov 2. PMID 22056301